CLINICAL TRIAL: NCT05509049
Title: Employing Machine Learning and Behavioral Science Solutions to Increase Women's Wellness Scheduling and Attendance: A Randomized Controlled Trial
Brief Title: Precision Nudging Drives Wellness Visit Attendance at Scale
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lirio (Industry)
Collaborators: Rochester Regional Health (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: LRRHWWRCT; IRB 2129 (Other: Rochester Regional Health Institutional Review Board)
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Women's Health; Annual Visit; Well Visit; Health Behavior; Prevention
Keywords: Digital Health Intervention; Behavior Change; Reinforcement Learning; Artificial Intelligence
MeSH Terms: conditions — Health Behavior | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective, parallel, large simple superiority randomized controlled trial using simple randomization (no blocking, no stratification).
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Behavioral science and reinforcement learning-driven hyper-personalized messages
  Interventions: Other: Precision nudging
- Control (Active Comparator): Standard of care message
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Precision nudging — Precision nudging (i.e., the application of behavioral science and reinforcement learning to create individualized, tailored health messaging at scale that matches the right message to the right person at the right time)
  Arms: Treatment
Other: Standard of care — Standard of care communication (e.g., personalized letters and patient portal notices)
  Arms: Control

SUMMARY:
The purpose of the present randomized controlled trial is to explore the effectiveness of a 12-month well woman digital health intervention leveraging Precision Nudging - the application of behavioral science and reinforcement learning to create individualized, tailored health messaging at scale that matches the right message to the right person at the right time - in promoting behavior change. Specifically, it is hypothesized that scaling behavioral science through reinforcement learning will be more effective at motivating participants to engage with well woman messages and to schedule and to attend a well woman visit compared to a standard of care message.

ELIGIBILITY:
Inclusion Criteria:

* Patient of health care system.
* Visit with OBGYN office in the last 36 months.
* OBGYN office provider is a Women's Wellness group approved provider.

Exclusion Criteria:

* Completed a women's wellness within the last 366 days.
* Upcoming women's wellness appointment.
* Had a childbirth episode (e.g., C-section vaginal delivery, or other event, including stillbirth) within the last 3 months or has a pregnancy due date in the future.
* Unsubscribed.

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30068 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who attended a well woman visit | 3 months
Proportion of participants who attended a well woman visit | 6 months
Proportion of participants who attended a well woman visit | 9 months
Proportion of participants who attended a well woman visit | 12 months
Proportion of participants who scheduled a well woman visit | 3 months
Proportion of participants who scheduled a well woman visit | 6 months
Proportion of participants who scheduled a well woman visit | 9 months
Proportion of participants who scheduled a well woman visit | 12 months
Proportion of participants who scheduled a well woman visit and did not attend (and did not Cancel and/or Reschedule) | 3 months
Proportion of participants who scheduled a well woman visit and did not attend (and did not Cancel and/or Reschedule) | 6 months
Proportion of participants who scheduled a well woman visit and did not attend (and did not Cancel and/or Reschedule) | 9 months
Proportion of participants who scheduled a well woman visit and did not attend (and did not Cancel and/or Reschedule) | 12 months

SECONDARY OUTCOMES:
Proportion of participants who opened and/or clicked Call-to-Action, or otherwise engaged with the communication(s) | 3 months
Proportion of participants who opened and/or clicked Call-to-Action, or otherwise engaged with the communication(s) | 6 months
Proportion of participants who opened and/or clicked Call-to-Action, or otherwise engaged with the communication(s) | 9 months
Proportion of participants who opened and/or clicked Call-to-Action, or otherwise engaged with the communication(s) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Ernest, DNP, BSN, MS, WHNP-C, Principal Investigator — Rochester Regional Health
Locations (1):
- Rochester Regional Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No